CLINICAL TRIAL: NCT01759134
Title: Comparison of Post-Discharge Growth of Premature Infants Using Two Different Formulas
Status: Terminated | Phase: Phase 4 | Type: Interventional
Sponsor: Shaare Zedek Medical Center (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: chammermanpdc
Record Dates: First submitted 2012-01-02; First posted 2013-01-02 (Estimated); Last update posted 2013-10-25 (Estimated); Status verified 2012-12

CONDITIONS: Premature Birth of Newborn
Keywords: Premature neonate; Post-discharge; Formula
MeSH Terms: conditions — Premature Birth

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Post Discharge Formula (Experimental): Babies will be given formula for first three months post discharge
  Interventions: Other: Post discharge formula

INTERVENTIONS:
Other: Post discharge formula — Babies will be given either materna sensitive or similac neosure

SUMMARY:
The objective of this study is to compare the post-discharge growth of preterm infants fed with 2 different post discharge formulas.

DETAILED DESCRIPTION:
Infants will be randomized upon discharge from the NICU. We will follow weight, height and head circumference for three months following discharge, In addition any feeding difficulties will be noted.

ELIGIBILITY:
Inclusion Criteria:

1. Preterm infants that are being fed only by formulas (mother chose not to breast feed, or cannot breast feed).
2. Gestational week 30-34.

Exclusion Criteria:

1. Congenital major malformation (e.g. congenital heart disease).
2. Chromosomal abnormality (e.g. Down's syndrome)
3. Gastrointestinal morbidity: S/P abdominal surgery, S/P NEC
4. Milk allergy
5. Chronic disease (e.g. oxygen treatment)

Ages: 30 Weeks to 34 Weeks | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 30 (Estimated)
Dates: Start 2013-01; Primary Completion 2014-01 (Estimated); Study Completion 2014-06 (Estimated)

PRIMARY OUTCOMES:
growth | 3 months post discharge
  weight (kg), length (cm), head circumference (cm).

CONTACTS AND LOCATIONS:
Overall Officials: Alona Bin-Nun, MD, Principal Investigator — Shaare Zedek Medical Center; Cathy Hammerman, MD, Principal Investigator — Shaare Zedek Medical Center
Locations (1):
- Shaare Zedek Medical Center, Jerusalem, Israel